CLINICAL TRIAL: NCT06551792
Title: The Effect of Magnesium Deficiency on Transforaminal Epidural Steroid Injection Success: An Observational Study
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Halil Ibrahim Altun, pain specialist, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: KanuniSS
Record Dates: First submitted 2024-04-24; First posted 2024-08-13 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Pain, Back
Keywords: pain,magnesium level, disc herniation
MeSH Terms: conditions — Back Pain; Intervertebral Disc Displacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Effect of Serum Magnesium Level on the Success of Transforaminal Epidural Steroid Injection: Transforaminal Epidural Steroid Injection groups
  Interventions: Other: Effect of Serum Magnesium Level on the Success of Transforaminal Epidural Steroid Injection

INTERVENTIONS:
Other: Effect of Serum Magnesium Level on the Success of Transforaminal Epidural Steroid Injection — Effect of Serum Magnesium Level on the Success of Transforaminal Epidural Steroid Injection

SUMMARY:
Transforaminal epidural steroid injection (TFESE) is an interventional method frequently used in the treatment of radicular pain due to disc herniation. TFESE, which is applied under sterile conditions and under fluoroscopy guidance, increases its effectiveness when applied in the early period (first 3 months). Inflammation and increase in neurotransmitters in the nerve root due to disc herniation trigger pain. Steroids and local anesthetics applied to the nerve root with TFESE exhibit strong anti-inflammatory effects. Factors affecting the success of TFESE include the type and dose of drugs, the age of the patient, any accompanying comorbidities, the level of injection administered and other musculoskeletal problems. Studies on the effect of these parameters on the effectiveness of TFESE are limited.Cardiac arrhythmia, muscle spasms, tetany, fasciculation paresthesia, widespread body pain, impaired bone mineralization, electrolyte disorders such as hypokalemia, hypocalcemia, hypophosphatemia, depression, and seizures may occur due to magnesium deficiency. One of the most important causes of low back pain is degenerative disc disease, and magnesium deficiency has been shown to be associated with low back pain.

DETAILED DESCRIPTION:
The study will be conducted by retrospectively scanning the files of patients with paracentral/subarticular protruded disc herniation and who underwent transforaminal epidural steroid injection (TFESE) to the lumbosacral region, at the Algology Department of Kanuni Sultan Süleyman Training and Research Hospital, between January 2022 and January 2024. In order to prevent heterogeneity, magnetic resonance imaging (MRI) of the patients will be evaluated in consultation with a radiologist. The common consensus classification created by the American Society of Spine Radiology (ASSR), American Society of Neuroradiology (ASNR) and North American Spine Society (NASS) is used to classify disc herniations. will be used. Numeric Rating Scale-11 (NRS) and Oswestry Disability Index (ODI) will be recorded from the patients' files before the procedure, in the first month and in the third month to evaluate age, gender, symptom duration, pain and functionality. The initial pain severity of the patients will be determined by the NRS-11 score, and a decrease of 50% or more in the NRS-11 score in the first month after the procedure will be considered as benefiting from the treatment. The Mg level of the patients before the procedure will be scanned in the hospital system and those that can be accessed will be recorded.

ELIGIBILITY:
Exclusion Criteria:

* Patients whose medical analgesic treatment was changed during their three-month follow-up;
* Those with fibromyalgia;
* Those with metabolic diseases (chronic renal failure, spondyloarthropathies, diabetes, hypo/hyperthyroidism, etc.) that may affect serum magnesium level;
* Those with a history of lumbar surgery;
* those taking magnesium or calcium supplements;
* Those with malignancy or obesity;
* Those with psychiatric illness;
* Those without lumbar MRI; Patients whose clinical, physical examination and laboratory data cannot be accessed

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusion Criteria:
  * Patients with paracentral/subarticular protruded disc herniation who underwent transforaminal epidural steroid injection (TFESE) to the lumbosacral region
  * Patients with complete data to be scanned in their files
Sampling Method: Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale-11 (NRS-11) | 3 months
  It is an 11-point scale used to describe pain. It is based solely on the patient ability to perform activities of daily living and can be used for adults and children ages 10 and older.

SECONDARY OUTCOMES:
Oswestry Disability Index | 3 months
  The self-completed questionnaire contains ten topics concerning intensity of pain, lifting, ability to care for oneself, ability to walk, ability to sit, sexual function, ability to stand, social life, sleep quality, and ability to travel.

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni Sultan Süleyman Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No